CLINICAL TRIAL: NCT00295776
Title: Lamictal in the Treatment of Post-Herpetic Neuralgia-A Safety, Efficacy,Randomized, Double Blind, Placebo Controlled, Cross-Over Study
Brief Title: Lamictal in the Treatment of Post-Herpetic Neuralgia
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: enrollment difficult due to inclusion/exclusion criteria/protocol requirements
Sponsor: George Washington University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: Lamictal PHN
Record Dates: First submitted 2006-02-22; First posted 2006-02-24 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2005-02

CONDITIONS: Neuralgia, Postherpetic
Keywords: Inclusion Criteria:Minimum of 4 on the Likert Pain Scale.If currently taking TCA and/or Gabapentin, need to have been on stable dose for minimum of 4 weeks.; Exclusion Criteria:; Currently on any antiepilepic drugs (AED), except for Gabapentin.; Currently taking opioid or unwilling to washout prior to the study,; Pregnant and lactating,; Have active severe systemic disease,; History of Stevens-Johnson syndrome or TEN,
MeSH Terms: conditions — Neuralgia, Postherpetic; Stevens-Johnson Syndrome | interventions — Lamotrigine

INTERVENTIONS:
Drug: Lamictal in the treatment of Post-Herpetic Neuralgia

SUMMARY:
To assess the efficacy of Lamictal for the treatment of pain and reduction of allodynia in patients with post herpetic neuralgia.

ELIGIBILITY:
Inclusion Criteria:

* All patients will be over the age of 18,
* Need to have a diagnosis of Post-Herpetic Neuralgia,
* Minimum of 4 on the Likert Pain Scale,
* If currently taking TCA and/or Gabapentin, need to have been on stable dose for minimum of 4 weeks

Exclusion Criteria:

* Currently on any antiepileptic drugs (AED), except for Gabapentin.
* Currently taking opioid or unwilling to washout prior to the study,
* Pregnant and lactating,
* Have active severe systemic disease,
* History of Stevens-Johnson syndrome or TEN,
* Clinically significant abnormal lab values,
* Known drug allergy to Lamictal,
* Patients on Fibrates (Tricor and Lopid),
* History of major psychiatric disturbance and substance abuse.
* Valproate due to increase chances of severe rash,
* Lidocaine Patch,
* Use of hormonal contraceptives (birth control pills, patch, ring, injection)

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2005-02; Primary Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Perry K. Richardson, M.D., Principal Investigator — The George Washington University Medical Faculty Associates
Locations (1):
- Medical Faculty Associates, Washington D.C., District of Columbia, United States